CLINICAL TRIAL: NCT02278978
Title: A Phase II Trial of BIBF1120 in Patients With Advanced FGFR3 Mutated, FGFR3 Overexpressed, or FGFR3 Wild Type Urothelial Carcinoma of Urinary Bladder, Urethra, Ureter, and Renal Pelvis and Who Have Failed Platinum-based Chemotherapy
Brief Title: BIBF1120 in Patients With Advanced FGFR3 Mutated,Overexpressed,or Wild Type Urothelial Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201306022MIPB
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Urothelial Carcinoma
Keywords: urothelial carcinoma; BIBF1120
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- FGFR3 mutated (Experimental): BIBF 1120 in patients with advanced FGFR3 mutated
  Interventions: Drug: BIBF1120
- FGFR3 overexpressed (Experimental): BIBF 1120 in patients with advanced FGFR3 overexpressed
  Interventions: Drug: BIBF1120
- FGFR3 wild type (Experimental): BIBF 1120 in patients with advanced FGFR3 wild type
  Interventions: Drug: BIBF1120

INTERVENTIONS:
Drug: BIBF1120 — BIBF1120 200 mg two times per day orally
  Other Names: Nintedanib

SUMMARY:
BIBF1120 in patients with advanced FGFR3 mutated, FGFR3 overexpressed, or FGFR3 wild type urothelial carcinoma of urinary bladder, urethra, ureter, and renal pelvis and who have failed platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* KPS 60%
* Histological confirmation of urothelial carcinoma , with metastatic disease
* Measurable disease
* Previously treated with platinum-based chemotherapy administered

Exclusion Criteria:

* Radiographic evidence of cavitary or necrotic tumours
* Active brain metastasis.Leptomeningeal metastasis
* Chemotherapy, radiotherapy, targeted therapy with monoclonal antibodies or small tyrosine kinase inhibitors
* Grade 1 treatment-related toxicity from previous chemotherapy, radiotherapy, or targeted therapy
* Prior treatment with BIBF 1120 or other VEGFR inhibitors
* Significant cardiovascular diseases:
* Pericardial effusion
* Significant bleeding or thrombosis
* Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug
* Major injuries within the past 10 days with incomplete wound healing and/or planned surgery during the on-treatment study period

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Response rate assessed by RECEST version 1.1 | 2 months
  To define the response rate of BIBF1120 in patients with advanced FGFR3-mutated,overexpressed,wild type UC and who have failed platinum-based chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Chi Lin, Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Chia-Chi Lin, Taipei, Taiwan